CLINICAL TRIAL: NCT01400360
Title: Invasive Diagnostic and Therapeutic Management of Cerebral Vasospasm After Aneurysmatic Subarachnoid Hemorrhage
Acronym: IMCVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Hartmut Vatter, M.D., Dept. of Neurosurgery, Goethe-University Frankfurt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JohannWGUH_IMCVS
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-05

CONDITIONS: Cerebral Vasospasm After Subarachnoid Hemorrhage
Keywords: cerebral vasospasm; subarachnoid hemorrhage; transluminal balloon angioplasty; intraarterial treatment
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- invasive (Active Comparator): After proof of perfusion relevant CVS in interventional therapy should be performed as best possible combination from TBA and intraarterial vasodilators additional to the conventional treatment.
  Interventions: Other: Combination of TBA and intraarterial application of vasodilators
- conventional (No Intervention): After proof of perfusion relevant CVS only conventional treatment should be performed (no intraarterial therapy).
  Interventions: Other: Combination of TBA and intraarterial application of vasodilators

INTERVENTIONS:
Other: Combination of TBA and intraarterial application of vasodilators — In the invasive arm CVS should be treated by intraarterial therapy and efficacy controlled by CT or MRI after 48 hours and if necessary repeated.

SUMMARY:
Cerebral vasospasm(CVS) after subarachnoid hemorrhage (SAH) results in a considerable amount of transient or even permanent neurological deficits and poor outcome of the patients. Transluminal Balloon angioplasty (TBA) or intraarterial application of vasodilators represents a rescue therapy for severe CVS. Indication, duration and efficacy of this treatment, however, is still under debate. Aim of the study is to investigate if such a rescue treatment can significantly reduce new delayed ischemic cerebral deficits after SAH. Hypothesis is that the occurance of delayed infarcts can be reduced by repetetive intraarterial therapy to more than 50 %.

ELIGIBILITY:
Inclusion Criteria:

* SAH (WFNS 1-4)
* Perfusion relevant CVS
* Ability for MRI, DSA and intraarterial treatment

Exclusion Criteria:

* extended cerebral infarcts
* SAH or ICH from AVM or flow associated aneurysm
* Non aneurismal SAH
* Relevant non spastic stenosis of brain supplying arteries

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
New infarcts between baseline and final MRI | 21 + - 7 days

SECONDARY OUTCOMES:
Clinical outcome (mRS, Karnofsky) | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Neurochirurgische Klinik, Universitätsklinik, Düsseldorf
  - Department of Neurosurgery, Johann Wolfgang Goethe-University, Frankfurt am Main
  - Neurochirurgische Klinik der Universität Ulm, Günzburg
  - Klinik für Neurochirurgie, Universitätsklinikum, Jena
  - Klinik für Neurochirurgie, Universitätsklinikum, Mannheim